CLINICAL TRIAL: NCT06383962
Title: A Single Site Post-Market Data Collection Protocol to Evaluate the Performance of Synergy Spine Solutions Synergy Disc®
Brief Title: Post-Market Data Collection to Evaluate the Performance of the Synergy Disc®
Status: Recruiting | Type: Observational
Sponsor: Synergy Spine Solutions (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: CP 21-001-UK02
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cervical Degenerative Disc Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective: All patients for whom the decision has been made to have the Synergy Disc system implanted and give informed consent will be enrolled in this study, following country-specific requirements.
  Interventions: Device: Synergy cervical spine disc replacement
- Retrospective: Patients who have previously received the Synergy Disc system in the last ten years are eligible for inclusion in the retrospective data collection; a waiver of consent, or an informed consent, for the retrospective data collection from the medical records of the implanting surgeon will be sought per country-specific regulations.
  Interventions: Device: Synergy cervical spine disc replacement

INTERVENTIONS:
Device: Synergy cervical spine disc replacement — motion preservation disc

SUMMARY:
This is a real world data collection observational study at a single site. There are both prospective and retrospective cohorts. The study will examine the safety and effectiveness of the Synergy cervical disc system in patients with degenerative cervical disc disease.

ELIGIBILITY:
Inclusion Criteria:

Age 21 or above at the time of the surgery. Have had (retrospective cohort) or the decision has been made to have (prospective cohort) the Synergy Disc implanted Skeletally mature patients for reconstruction of the disc from C3-C7 following a single or multiple level discectomy for intractable radiculopathy

Intractable radiculopathy and/or myelopathy with at least one of the following producing symptomatic nerve root and/or spinal cord compression:

herniated disc and/or osteophyte formation Symptomatic nerve root and/or spinal cord compression documented by patient history (arm or neck pain and/or neurologic deficit) and imaging (CT, MRI, x-rays, etc.) Failed a minimum of 6 weeks conservative treatment Written informed consent given by subject.

Exclusion Criteria:

Exclusion Criteria: All answers must be NO to be eligible for the study. Moderate to advanced spondylosis Diagnosis of osteoporosis Active systemic infection or infection at the operative site Pregnancy Marked cervical instability on lateral, coronal, or flexion/extension radiographs Cervical spine condition other than symptomatic cervical disc disease requiring surgical treatment at the involved level Severe pathology of the facet joints of the involved vertebral bodies Previous diagnosis of osteopenia or osteomalacia More than one immobile vertebral level between C1 and T1 from any cause Morbid obesity Vulnerable person (pregnant patients, emergency cases, children, prisoners and people without mental capacity)

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who have had (retrospective cohort) or who are going to (prospective cohort) the Synergy cervical disc and have cervical degenerative disc disease that has been unresponsive to conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | 12 months
  Neck disability Index improvement of >15 pts (out of 100) in subjects by 12 months post operative compared with baseline. A lower score is a better score.
Device Related or Device Procedure Related Adverse Events | 12 months
  Absence of major device related adverse events defined as radiographic failure, neurologic failure or failure by adverse event

SECONDARY OUTCOMES:
Neck and Arm Pain Measurement | pre-operative, 6 week, 3 month, 6 month, 12 month, 24 month
  Pain will evaluated by the Visual analog scale (VAS) (place a line from zero where there is no pain to 10 which is the worst pain imaginable), by NRS (circle a number from zero to ten where zero equals no pain and ten is worst imaginable) to or a verbal description that the doctor writes down, per the site's Standard of Care. A change of at least 20 mm will be considered clinically significant. Neck pain as measured on a 100mm VAS at baseline and at each follow-up timepoint. Left and Right arm/shoulder pain as measured on a 100 mm VAS at baseline and at each follow up time-point.
Patient Satisfaction | 6 week, 3 month, 6 month, 12 month, 24 month
  patient completed questionnaire on their satisfaction with the disc replacement surgery
Motor and Sensory Function in the Arm | pre-operative, 6 week, 3 month, 6 month, 12 month, 24 month
  maintenance or improvement in neurologic status compared with baseline will be assessed using a defined numeric scale ranging from 0 (normal) to 5 (deficit)
Nurick's Criteria | pre-operative, 6 week, 3 month, 6 month, 12 month, 24 month
  Disease status as characterized by physician at each time point
Odom's criteria | pre-operative, 6 week, 3 month, 6 month, 12 month, 24 month
  surgical outcome characterized by physician at each post operative visit

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Capobianco, PhD, Study Director — Synergy Spine Solutions
Locations (2):
- United Kingdom (2):
  - Royal Orthopaedic Hospital, Birmingham
  - Kings College Hospital, London

IPD SHARING:
Plan to Share IPD: No